CLINICAL TRIAL: NCT04993040
Title: A Clinical Study to Determine the Pharmacokinetics of Oraxol in Breast Cancer Patients
Brief Title: A PK Study of Oraxol in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-CN-007
Record Dates: First submitted 2019-03-11; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-02

CONDITIONS: Breastcancer
Keywords: breast cancer; paclitaxel
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oraxol (Experimental): Subjects will receive Oraxol 205 mg/m2 daily x 3 days weekly for up to 16 weeks.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — * HM30181 methanesulfonate monohydrate
  * Oral paclitaxel capsules
  Other Names: HM30181 methanesulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets, Paclitaxel - supplied as 30-mg capsules

SUMMARY:
This is a multicenter, open-label, single-arm PK study in approximately 24 breast cancer patients for whom paclitaxel treatment is indicated.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm PK study in approximately 24 breast cancer patients for whom paclitaxel treatment is indicated. The study contains 3 periods: the Screening / Baseline Period, the Treatment Period, and the Follow-up Period. A Final Visit will occur within 7 days of the last dose of study treatment. If subjects achieve stable disease (SD), partial response (PR), or complete response (CR) at the end of the Treatment Period, they may continue Oraxol treatment in a separate extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Women ≥18 years of age on day of consent
3. Breast cancer in patients for whom treatment with IV paclitaxel at 80 mg/m2 as monotherapy has been recommended by their oncologist.
4. Measurable disease as per RECIST v1.1 criteria
5. Adequate hematological status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Hemoglobin (Hgb) ≥9 g/dL
6. Adequate liver function as demonstrated by:

   * Total bilirubin of ≤1.5 mg/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present
   * Alkaline phosphatase (ALP) ≤3 x ULN or ≤5 x ULN if bone metastasis is present
   * Gamma glutamyl transferase (GGT) <10 x ULN
7. Adequate renal function as demonstrated by serum creatinine ≤1.5 x ULN
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Life expectancy of at least 3 months
10. Willing to fast for 6 hours before and 2 hours after Oraxol administration on all treatment days
11. Willing to abstain from alcohol consumption for 3 days before the first dose of study drug through the completion of the second inpatient PK sampling period
12. Willing to refrain from caffeine consumption for 12 hours before each inpatient dosing period (Weeks 1 and 4) through the completion of protocol-specified PK sampling for that week
13. Subjects must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of assigned study treatment.
14. Subjects who are of childbearing potential must have a negative serum pregnancy test at Screening and within 96 hours before Week 1 dosing.

Exclusion Criteria:

1. Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products (IPs)
2. If previously treated with a taxane (paclitaxel or docetaxel) as part of anthracycline-based adjuvant chemotherapy or for metastatic disease, the subject relapsed less than 1 year following treatment
3. Subjects unable to swallow study medication in its intact form or have clinically significant malabsorption syndrome
4. Only site of metastatic disease is unmeasurable according to RECIST v1.1 criteria
5. Known CNS metastasis, including leptomeningeal involvement
6. Received IPs within 14 days or 5 half-lives of the first study dosing day, whichever is longer
7. Are currently receiving other medications intended for the treatment of their malignancy
8. Women who are pregnant or breastfeeding
9. Taking any of the following prohibited medications:

   * Strong inhibitors (eg, ketoconazole) or inducers (eg, rifampin or St. John's Wort) of CYP3A4 (within 2 weeks prior to the start of dosing in the study)
   * Strong inhibitors (eg, gemfibrozil) or inducers (eg, rifampin) of CYP2C8 (within 2 weeks prior to the start of dosing in the study)
   * Strong P-gp inhibitors or inducers. Subjects who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication ≥1 week before dosing and remain off that medication through the end of study treatment.
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg,digoxin, dabigatran) within 24 hours prior to start of dosing in the study
10. Use of warfarin. Subjects receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
12. Known allergic reaction or intolerance to study medication components
13. Known allergic reaction or intolerance to contrast media
14. Subjects who, in the Investigator's opinion, are not suitable for participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Cmax | Week 1 (Days 1,2, 3): Predose, and at 1, 2, 3, and 4 hours postdose; Week 4 (Days 1,2,3): Predose, and at 1, 2, 3, and 4 hours postdose
  Plasma concentrations for paclitaxel only will be analyzed to determine the maximum observed concentration (Cmax).
  Pharmacokinetic parameters will be summarized using the mean, standard deviation, median, minimum, and maximum. Summaries of PK parameters will also include the geometric mean and the coefficient of variation. Summary PK and individual timepoints will be tabulated and displayed graphically and listed for all subjects.
Cmin | Week 1 (Days 1,2, 3): Predose, and at 1, 2, 3, and 4 hours postdose; Week 4 (Days 1,2,3): Predose, and at 1, 2, 3, and 4 hours postdose
  Plasma concentrations for paclitaxel only will be analyzed to determine the minimum observed concentration (Cmin).
  Pharmacokinetic parameters will be summarized using the mean, standard deviation, median, minimum, and maximum. Summaries of PK parameters will also include the geometric mean and the coefficient of variation. Summary PK and individual timepoints will be tabulated and displayed graphically and listed for all subjects.
Cavg | Week 1 (Days 1,2, 3): Predose, and at 1, 2, 3, and 4 hours postdose; Week 4 (Days 1,2,3): Predose, and at 1, 2, 3, and 4 hours postdose
  Plasma concentrations for paclitaxel only will be analyzed to determine the area under the curve extrapolated to infinity (AUC0-t).
  Pharmacokinetic parameters will be summarized using the mean, standard deviation, median, minimum, and maximum. Summaries of PK parameters will also include the geometric mean and the coefficient of variation. Summary PK and individual timepoints will be tabulated and displayed graphically and listed for all subjects.
AUC0-t | Week 1 (Days 1,2, 3): Predose, and at 1, 2, 3, and 4 hours postdose; Week 4 (Days 1,2,3): Predose, and at 1, 2, 3, and 4 hours postdose
  Plasma concentrations for paclitaxel only will be analyzed to determine the area under the curve (AUC).
  Pharmacokinetic parameters will be summarized using the mean, standard deviation, median, minimum, and maximum. Summaries of PK parameters will also include the geometric mean and the coefficient of variation. Summary PK and individual timepoints will be tabulated and displayed graphically and listed for all subjects.
AUC | Week 1 (Days 1,2, 3): Predose, and at 1, 2, 3, and 4 hours postdose; Week 4 (Days 1,2,3): Predose, and at 1, 2, 3, and 4 hours postdose
  Plasma concentrations for paclitaxel only will be analyzed to determine the area under the curve (AUC).
  Pharmacokinetic parameters will be summarized using the mean, standard deviation, median, minimum, and maximum. Summaries of PK parameters will also include the geometric mean and the coefficient of variation. Summary PK and individual timepoints will be tabulated and displayed graphically and listed for all subjects.

SECONDARY OUTCOMES:
Safety | From screening until final visit (within within 7 days after last dose of study treatment)
  all AEs (including for both increasing and decreasing severity) and SAEs by CTCAE v4.03
Tumor response rate | From screening until final visit (within within 7 days after last dose of study treatment)
  which is defined as the number of subjects with complete response (CR) or partial response (PR) at any post-baseline assessments by RECIST 1.1
Progression-free survival | From date of dosing until the date of first documented progression or date of death from any cause, whichever came first, estimated up to 24 months
  Progression Free Survival (PFS) based on investigator's assessment according to RECIST 1.1
Overall survival | From date of dosing until the date of death from any cause, whichever came first, estimated up to 24 months
  OS is defined as the length of time from 1st dosing until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Pro.f, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Herui Yao, Pro.f, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided